CLINICAL TRIAL: NCT06977178
Title: Adverse Adolescent Pathways to Substance Use
Acronym: APSU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); RTI International (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-1572; 5R01DA057312-02 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Adolescent Development; Substance Use
MeSH Terms: conditions — Anxiety Disorders; Substance-Related Disorders | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: The Trier Social Stress Test for Children (TSST-C 61)-- a social stressor involving story telling in front of two neutral judges, preparation time and a cognitive stressor involving mental arithmetic-counting backward from 1023 by 13s--will be used to elicit physiological stress responses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trier Social Stress Test (TSST) (Experimental): The Trier Social Stress Test for Children (TSST-C) is a social stressor involving story telling in front of two neutral judges, preparation time and a cognitive stressor involving mental arithmetic-counting backward from 1023 by 13s. It is used to elicit physiological stress responses. The TSST-C is administered in 4 parts: an anticipatory stress phase (5 min to prepare the speech); the speech task (5 min), the arithmetic task (5 min), and the recovery phase (up through 40 min post-task).
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Psychosocial stress procedure; 5 minutes of public speaking (preceded by 5 minutes of preparation) and 5 minutes of mental arithmetic.

SUMMARY:
Purpose: This 5-year R01 study will elucidate the role of maturational change across adolescence in neural connectivity and physiological stress responses in the relationship between anxiety and adverse pathways to substance use (APSU). Participants: Children (N=200) aged 12-14 with symptoms of anxiety and their legal caregiver will be recruited from clinical and community sources. Procedures: Youth participants will complete several questionnaires and interviews, undergo neuroimaging while performing cognitive tasks, and have their heart rate and skin conductance monitored during a mildly stressful task. Caregivers will complete several questionnaires.

DETAILED DESCRIPTION:
The conceptual model proposes that the relationship between anxiety symptomatology and Adverse Patterns of Substance Use (APSU: age of onset, cumulative exposure, severity, and polydrug use) is a function of acute stress reactivity that is underpinned by specific neurobiological and neurocognitive factors measurable at a drug- and alcohol-naïve baseline. Youth at high risk for APSU will be over-sampled using parent and child-reported screeners that include items relating to emotion dysregulation, behavioral impulsivity, susceptibility to peer pressure, friends' conduct problems, and other risk-relevant characteristics to define a high-APSU-risk prodrome. Risk status will be measured as a continuous trait using well-tested thresholds for high and low risk for APSU, and the recruitment strategy will ensure sufficient variability on this axis. This approach ensures a sufficient number of youth will initiate and escalate SU within the time frame of the study, allowing the investigators to assess precursors APSU in high risk youth as a function of anxiety symptomatology and acute stress reactivity, using feasible and adequately powered methods.

To test hypotheses, the investigators will prospectively assess acute stress responsivity, anxiety symptoms, specific neural connectivity patterns, and APSU in a sample of 180 substance-naïve youth beginning in early adolescence (age 12-14, Tanner Stage >3) and two additional 12 month waves of data collection. Participants will complete an acute stress task outside the scanner with psychophysiological monitoring and a resting and performance based MRI session using impulsivity (fronto-striatal-thalamic circuitry), negative valence (threat circuitry), and attention bias (shifting from threat to frontal circuitry) tasks. At each wave, all surveys, cognitive tests, stress physiological, clinical and neuroimaging measures will be assessed. A final online exit survey in year 5 will be conducted simultaneously for all participants to evaluate clinical symptoms and end-point APSU.

The proposed prospective, longitudinal design is novel, creative, and timely. Brain imaging studies of this type are typically quite small, often due to cost limitations, and are only able to accurately model a small subset of factors and covariates. The investigators plan to evaluate the complexity of the problem with targeted variables that will be well-defined in the sample and tracked over time in relation to APSU in an atypically large sample for neuroimaging. This design will enable within- and between-subject comparisons that prospectively: (1) characterize substance use pathways (e.g., nature and extent of use over time) in the context of neurobiological and neurocognitive mechanisms associated with physiological responses to acute stress that underlie anxiety symptoms, (2) tracks developmental change in these processes, and (3) differentiates between potentially distinctive neural pathways that influence progression to APSU.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 12-14 years old,
* Report symptoms of anxiety
* Understand and sign an assent, and parents will sign a permission and a consent document in English
* Meets study hearing and vision requirements
* Substance use naïve

Exclusion Criteria:

* Has any foreign metal objects or implants as determined by the safety questionnaires (e.g., bone screws, shunts or body piercing that can't be removed, etc.)
* Has been diagnosed with psychosis or a severe emotional disturbance.
* Has used alcohol, tobacco, or marijuana more than 3 times.
* Is pregnant. Girls who self-report pregnancy may not participate in the stress evaluation or the MRI scan.
* Is taking any medications that directly alter cardiovascular function (e.g., propranolol or other beta blockers).
* Any current or lifetime treatment with antipsychotic medication.
* Has had a head injury that resulted in a loss of consciousness for more than 5 minutes.
* Is planning to get non-removable metal braces.
* Impaired intellectual functioning (full-scale intelligence quotient <70).
* Past or current history of a clinically significant central nervous system that could confound brain imaging evaluations.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Reaction time during the functional magnetic resonance imaging (FMRI) Stop Signal Task | baseline, 12-months, 24-months
  The Stop Signal Task is a measure of inhibitory control. Participants are presented with a right or left arrow and instructed to press one of two buttons corresponding with each arrow after it is presented. However, on certain trials, there is an up facing arrow immediately following the presentation of a left or right arrow, and participants are instructed to not press any buttons if they see an up arrow. The task measures the mean go reaction time to evaluate the participant's ability to inhibit when the up arrow is presented, with faster reaction times (measured in milliseconds) meaning lower inhibition.
Percent signal change during the FMRI Stop Signal Task | baseline, 12-months, 24-months
  Neural activation during the Stop Signal Task is measured through determining the percent signal change from baseline FMRI resting state to neural activation during the Stop Signal Task, particularly in the front-striatal-thalamic regions. Higher percent signal change would indicate higher levels of activation during the task. Percent signal change ranges between 1% to 5%.
Percent signal change activation during the No-stimuli, Predictable-stimuli, and Unpredictable-stimuli (NPU) task | baseline, 12-months, 24-months
  In the NPU task, participants are presented with fearful and neutral faces, with the fearful face presentation being sometimes cued with another associated visual stimuli immediately beforehand, and sometimes uncued and therefore unpredicted. This task measures cued anticipation of threat. The regions of interest are the intra-limbic regions, bed nucleus of the stria terminalis (BNST), and the amygdala. Higher percent signal change in these regions would indicate higher levels of activation during the task. Percent signal change ranges between 1% to 5%.
Percent signal change during the Attentional Load Paradigm (ALP) task | baseline, 12-months, 24-months
  In the ALP task, participants complete a letter search task while being presented with peripheral distractor letters on top of both fearful and neutral faces to evaluate the impact of perceptual load on the neural response to fearful vs neutral face distractors. The percent signal change will be specifically analyzed in the parietal and frontal cortices. Higher percent signal change in these regions would indicate higher levels of activation during the task. In addition, the ability to shift from affective-limbic to cognitive-pre-frontal cortex to complete the task will be evaluated as a key indicator of neural maturity. Percent signal change ranges between 1% to 5%.
Percent signal change during Emotional Face N-Back (EFNBack) | baseline, 12-months, 24-months
  In the EFNBack task, participants are shown images of emotionally salient (happy and fearful) and neutral faces as well as images of neutral places. Participants are instructed to determine whether each picture presented is a "Match" or a "No match". In the 0-back, low load condition, the "match" occurs when the picture presented is the same as a fixed target picture presented at the beginning. In the 2-back, high load condition, the "match" occurs when the picture presented is the same as the one shown two pictures ago. This task evaluates working memory and emotional regulation, as well as the percent signal change of the prefrontal cortex (PFC), amygdala, and anterior cingulate cortex (ACC), with higher percent signal change in these regions indicating higher levels of activation during the task. Percent signal change ranges between 1% to 5%.
Sympathetic and Parasympathetic nervous system ECG activation or heart rate variability (HRV) during a psychosocial stressful task (Trier Social Stress Test - TSST) | at baseline, 12-month and 24-month
  The Trier Social Stress Test for Children (TSST-C) -- a social stressor involving story telling in front of two neutral judges, preparation time and a cognitive stressor involving mental arithmetic-counting backward from 1023 by 13s -- is used to elicit physiological stress responses. The combination of stressors offers high levels of social-evaluative threat. The TSST-C will be administered in 4 parts: an anticipatory stress phase (5 min to prepare the speech); the speech task (5 min), the arithmetic task (5 min), and the recovery phase (up through 40 min post-task). For a five minute baseline period, and for the duration of the task, heart rate is measured to determine baseline resting state and HRV. HRV is the difference in the milliseconds between each heart beat. The higher the HRV, the more the nervous system is activated during the task. The level of HRV indicates the participant's nervous system response to stress.
Endocrine (cortisol) measures during a psychosocial stressful task (Trier Social Stress Test - TSST) | at baseline, 12-month and 24-month
  The Trier Social Stress Test for Children (TSST-C) -- a social stressor involving story telling in front of two neutral judges, preparation time and a cognitive stressor involving mental arithmetic-counting backward from 1023 by 13s-- is used to elicit physiological stress responses. The combination of these stressors offers elements of uncontrollability and high levels of social-evaluative threat. The TSST-C will be administered in 4 parts: an anticipatory stress phase (5 min to prepare the speech); the speech task (5 min), the arithmetic task (5 min), and the recovery phase (up through 40 min post-task). At rest, cortisol is collected through a saliva sample of passive drool. Then cortisol will be collected in 15 minute intervals for the duration of the task and recovery time. The higher the cortisol is found to be, the higher the stress response to the task.
Assessment of Liability and Exposure to Substance Use and Antisocial Behavior, Revised (ALEXSA-R) | at baseline, 12-month and 24-month
  The Assessment of Liability and Exposure to Substance use and Antisocial behavior, Revised (ALEXSA-R) is a system of youth-report measures of risks, resiliencies, risky health behavior. The youth-report Youth Risk Index (YRI) which is part of the ALEXSA-R will be used to screen for participants who are at high and low risk for early- to mid-adolescent problematic substance use. The YRI screening tool is designed for well-child visits to identify at-risk youths and refer them for prevention. The higher the YRI score (range 0-3) the higher the youth risk level.
Neurocognitive testing and executive functioning through NIH Toolbox | at baseline, 12-month and 24-month
  Neurodevelopmental maturity and cognitive functioning will be evaluated with NIH Cognitive Toolbox - Child Computerized performance tasks. These tasks test decision making, impulsivity, working memory, and attention. There is a memory task involving remembering the sequence of words, there is an inhibitory task involving pressing only certain buttons, and an attention task involving determining which pictures match and which do not. Each task produces a t score, with higher scores indicating higher performance on each task.
Multidimensional Anxiety Scale for Children 2 (MASC2) | at baseline, 12-month and 24-month
  The MASC2 is a comprehensive assessment of anxiety. It is a self-report scale for youth ages 8-19 with 50 items. It measures symptom severity, as well as range of symptoms across possible anxiety disorders and produces a t score which represents anxiety severity. This score can range from less than 40 (a low score) to above 70 (a high score).
State-Trait Anxiety Inventory for Children (STAI-C) | at baseline, 12-month and 24-month
  The STAI-C is a measure with two sub-surveys, with each one having 20 items each. The State measure assesses current anxiety at the moment of assessment, with a higher score meaning higher current anxiety. The Trait measure assesses level of anxiety severity in general as a trait of the participant, with a higher score meaning higher overall anxiety. The range in scores is between 20-80 for each sub-survey.
Tobacco Alcohol and Drug Use Survey | 12-month and 24-month
  Self-report survey to assess the frequency of use of multiple drugs: e.g., tobacco, alcohol, marijuana, cocaine, methamphetamine, opioids, etc. as the primary initial tool to assess what substances have been used by participants. This measure produces the number of days in the past year that the participant has used a substance as well as how recently the participant has used a substance.

SECONDARY OUTCOMES:
Age | at baseline, 12-month and 24-month
  Participant age is used as a secondary outcome to determine the impact of age on the primary outcome measures. Participant age falls in the range of 12-17.
Adverse Life Experiences | at baseline, 12-month and 24-month
  The Adverse Life Experiences Scale (ALES) is used to assess experiences of adversity, abuse, neglect, and threat. It will be used as a secondary outcome to determine the impact of adverse life experiences on the primary outcome measures. The number of adverse experiences reported by each participant is totaled, with the higher number of experiences meaning a higher level of adversity.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenil Belger, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the federal funding for this grant, participant's de-identified data will be uploaded to the NIMH data archive. The NIH-funded research data repository aims to accelerate progress in clinical research through data sharing, data harmonization, and the reporting of research results. It also serves as a scientific community platform and portal to multiple other research repositories, allowing for aggregation and secondary analysis of data. NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental health problems to collect and share de-identified information with each other.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available by 18 months past the study completion date. After uploading, the data will be available in the NDA long term, but must be kept on the NDA for at least three years after the funding period ends.
Access Criteria: De-identified data will be submitted to the National Institute of Mental Health Data Archive (NDA). To obtain access to the NDA, researchers follow the established procedures within NDA, and the NDA Data Access Committee will determine the approvals for these requests. Access will be given for any legitimate scientific purpose, as determined by NDA Access Committee.
URL: https://nda.nih.gov/